CLINICAL TRIAL: NCT02976753
Title: 24-month Prospective, Multicentre, Non-interventional Study to Evaluate the Effectiveness of Elocta Compared to Conventional Factor Products in the Prophylactic Treatment of Patients With Haemophilia A (A-SURE)
Brief Title: Prospective, Non-interventional Study to Evaluate the Effectiveness of Elocta Compared to Conventional Factor Products
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.Elocta-002
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Hemophilia A
Keywords: Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn
MeSH Terms: conditions — Hemophilia A; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — factor VIII-Fc fusion protein; Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Elocta: Elocta will be prescribed and administered for prophylactic treatment of patients with haemophilia A according to usual clinical practice
  Interventions: Drug: efmoroctocog alfa
- Conventional factor VIII product: Conventional factor VIII products will be prescribed and administered for prophylactic treatment of patients with haemophilia A according to usual clinical practice
  Interventions: Drug: Factor VIII

INTERVENTIONS:
Drug: efmoroctocog alfa — extended half-life factor VIII product
  Other Names: Elocta
  Groups: Elocta
Drug: Factor VIII — conventional factor VIII product
  Groups: Conventional factor VIII product

SUMMARY:
The purpose of the study is to evaluate the effectiveness of Elocta compared to conventional factor products in the prophylactic treatment of patients with haemophilia A over a 24-month prospective period. Data will also be collected for a 12 month retrospective period.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with a diagnosis of haemophilia A
* Received prophylactic treatment with a factor product for management of haemophilia A in the 12 months prior to enrolment
* At enrolment prescribed prophylactic treatment with Elocta or conventional factor product regardless of participation in the study
* Having at least 12 months documented pre-study treatment data regarding prophylactic treatment prescriptions and bleeding episodes prior to the baseline visit
* Signed and dated informed consent provided by the patient or the patient's legally acceptable representative for patients under the legal age before any study-related activities are undertaken. Assent should be obtained from paediatric patients according to local regulations

Exclusion Criteria:

* Enrolment in a concurrent clinical interventional study involving intake of an investigational medicinal product (IMP), within 1 year prior to enrolment
* Previously treated with commercially available extended half-life products other than Elocta
* Presence of factor VIII inhibitors (≥0.60 Bethesda Unit [BU]/mL ) at the latest available inhibitor test using the Nijmegen modified Bethesda assay

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male patients with a diagnosis of haemophilia A prescribed prophylactic treatment with Elocta or conventional factor product
Sampling Method: Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Annualised bleeding rate (ABR) | 24 months
Annualised injection frequency | 24 months
Annualised factor consumption (International Unit [IU]) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, MD, Study Director — Sweden Orphan Biovitrum
Locations (36):
- Austria (4):
  - Swedish Orphan Biovitrum Research site, Innsbruck
  - Swedish Orphan Biovitrum Research site, Linz
  - Swedish Orphan Biovitrum Research Site, Sankt Pölten
  - Swedish Orphan Biovitrum Research site, Vienna
- Swedish Orphan Biovitrum Research site, Brussels, Belgium
- Swedish Orphan Biovitrum Research site, Helsinki, Finland
- France (4):
  - Swedish Orphan Biovitrum Research site, Caen
  - Swedish Orphan Biovitrum Research site, Montpellier
  - Swedish Orphan Biovitrum Research site, Nancy
  - Swedish Orphan Biovitrum Research site, Rennes
- Italy (9):
  - Swedish Orphan Biovitrum Reserach site, Catanzaro
  - Swedish Orphan Biovitrum Reserach site, Florence
  - Swedish Orphan Biovitrum Research site, Milan
  - Swedish Orphan Biovitrum Reserach site, Naples
  - Swedish Orphan Biovitrum Research Site, Padua
  - Swedish Orphan Biovitrum Reserach site, Palermo
  - Swedish Orphan Biovitrum Reserach site, Parma
  - Swedish Orphan Biovitrum Reserach site, Rome
  - Swedish Orphan Biovitrum Research site, Turin
- Swedish Orphan Biovitrum Research site, Oslo, Norway
- Spain (6):
  - Swedish Orphan Biovitrum research site, Alicante
  - Swedish Orphan Biovitrum Reserach site, Barcelona
  - Swedish Orphan Biovitrum Reserach site, Madrid
  - Swedish Orphan Biovitrum Research site, Málaga
  - Swedish Orphan Biovitrum Reserach site, Seville
  - Swedish Orphan Biovitrum Research site, Valencia
- Sweden (3):
  - Swedish Orphan Biovitrum Research site, Gothenburg
  - Swedish Orphan Biovitrum Research site, Malmo
  - Swedish Orphan Biovitrum Research site, Stockholm
- United Kingdom (7):
  - Swedish Orphan Biovitrum Research site, Birmingham
  - Swedish Orphan Biovitrum Research site, Canterbury
  - Swedish Orphan Biovitrum Research site, Liverpool
  - Swedish Orphan Biovitrum Reserach site, London
  - Swedish Orphan Biovitrum Research site, Manchester
  - Swedish Orphan Biovitrum Research site, Sheffield
  - Swedish Orphan Biovitrum Research site, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oldenburg J, Hay C, Peyvandi F, Lehtinen AE, Pabinger I, Nuesch E, Malmstrom H, Bednar E, Lethagen S. A-SURE: intra-patient comparison of prophylactic effectiveness of a recombinant factor VIII Fc fusion protein versus standard half-life factor VIII in hemophilia A. Hematology. 2025 Dec;30(1):2513186. doi: 10.1080/16078454.2025.2513186. Epub 2025 Jul 4. PMID 40616274
- [Derived] Oldenburg J, Hay CRM, Jimenez-Yuste V, Peyvandi F, Schved JF, Szamosi J, Winding B, Lethagen S. Design of a prospective observational study on the effectiveness and real-world usage of recombinant factor VIII Fc (rFVIIIFc) compared with conventional products in haemophilia A: the A-SURE study. BMJ Open. 2019 May 30;9(5):e028012. doi: 10.1136/bmjopen-2018-028012. PMID 31152037